CLINICAL TRIAL: NCT06732713
Title: Effects Of Swiss Ball Versus Frenkel Exercises on Static and Dynamic Balance in Children With Down Syndrome.
Brief Title: Swiss Ball Versus Frenkel Exercises Effects in Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/24/0710
Record Dates: First submitted 2024-11-03; First posted 2024-12-13 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Swiss ball; Frenkel exercises; Static balance; Dynamic balance
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: The current study will be randomized clinical. The study will include 32 patients aged between 8 to 13 years equally divided into two groups and randomly allocated trial. Group A will perform Frenkel exercises and group B will perform Swiss ball exercises along routine physical therapy. Before and after intervention period, Static and dynamic balance will be assessed by Pediatric Balance Scale, Timed Up and Go test and Romberg test.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swiss ball group (Experimental): Swiss ball exercises will be done and intervention period will be of 8 weeks with 3 to 4 sessions per week of about 25 to 30 minutes
  Interventions: Other: Swiss Ball
- Frenkel exercise group (Experimental): Frenkel exercises will be done and intervention period will be of 8 weeks with 3 to 4 sessions per week of about 25 to 30 minutes
  Interventions: Other: Frenkel exercise

INTERVENTIONS:
Other: Swiss Ball — Swiss ball exercises will be performed in supine, sitting and standing position for about 25 to 30 minutes , 3 to 4 sessions per week for 8 weeks
  Arms: Swiss ball group
Other: Frenkel exercise — Frenkel exercises will be performed in supine, sitting and standing position for about 25 to 30 minutes, 3 to 4 sessions per week for 8 weeks
  Arms: Frenkel exercise group

SUMMARY:
Down syndrome (or trisomy 21) is the most common genetic cause of intellectual disability, occurring in an estimated 1 in 800 births worldwide. Approximately 11,000 people with Down syndrome live in Australia and 250,000 in the USA. Individuals with Down syndrome present with several impairments such as hypotonia, ligament laxity, decreased muscle strength, insufficient muscular co-contraction, inadequate postural control, and disturbed proprioception. Frenkel exercises are a series of motions of increasing difficulty performed by patients to facilitate the restoration of balance and coordination. Frenkel exercises are used to bring back the rhythmic, smooth and movements. In recent years, Swiss Ball has been widely used as a new method of treatment to increase balance, strengthen core region of body muscles, and strengthen muscles that are effective in maintaining posture, coordination, and flexibility. The aim of this recent study is to compare the effects of two different therapeutic techniques i.e Frenkel versus Swiss ball exercises on static and dynamic balance in children with Down syndrome.

DETAILED DESCRIPTION:
Down syndrome (or trisomy 21) is the most common genetic cause of intellectual disability, occurring in an estimated 1 in 800 births worldwide. Approximately 11,000 people with Down syndrome live in Australia and 250,000 in the USA. Individuals with Down syndrome present with several impairments such as hypotonia, ligament laxity, decreased muscle strength, insufficient muscular co-contraction, inadequate postural control, and disturbed proprioception. Frenkel exercises are a series of motions of increasing difficulty performed by patients to facilitate the restoration of balance and coordination. Frenkel exercises are used to bring back the rhythmic, smooth and movements. In recent years, Swiss Ball has been widely used as a new method of treatment to increase balance, strengthen core region of body muscles, and strengthen muscles that are effective in maintaining posture, coordination, and flexibility. The aim of this recent study is to compare the effects of two different therapeutic techniques i.e Frenkel versus Swiss ball exercises on static and dynamic balance in children with Down syndrome.

The current study will be randomized clinical trial, data will be collected from Children Hospital and Institute of Child Health, Lahore. The study will include 32 patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will include patients diagnosed with Down syndrome, age between 8 to 13 years, patient able to understand instructions necessary for intervention, independent standing and walking abilities. Patient with any heart deficit, visual or hearing disorder, mobility impairment and instability of atlanto occipital joint will be excluded. Sample will be divided into two groups.

Group A will perform Frenkel exercises and group B will perform Swiss ball exercises along routine physical therapy. Before and after intervention period, Static and dynamic balance will be assessed by Pediatric Balance Scale, Timed Up and Go test and Romberg test. Data collection will be done before and after the intervention. Data will be analyzed through SPSS version 23.00.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Down syndrome.
* Age between 8 to 13 years.
* Patient able to understand instructions necessary for intervention.
* Independent standing and walking abilities.
* Both the genders were included

Exclusion Criteria:

* Severe mental retardation.
* Any heart deficit.
* Visual impairments.
* Musculoskeletal or mobility disorder.
* Hearing impairements.
* Signs of epilepsy or instability of atlanto axial joint

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Pediatric Balance Scale | 8 weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Timed up and Go test | 8 weeks
  The 'timed up and go' test (TUG) is a simple, quick and widely used clinical performance- based measure of lower extremity function, mobility and fall risk.
  1. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
  2. On the word "Go," begin timing.
  3. Stop timing after patient sits back down.
  4. Record the time. The TUG has demonstrated good test-retest reliability (ICC 0.80-0.99), validity, and sensitivity to change. It has a moderate correlation with fall risk
Romberg test | 8 weeks
  Ask the subject to stand erect with feet together and eyes closed. Stand close by as a precaution in order to stop the person from falling over. Watch the movement of the body in relation to a perpendicular object behind the subject (corner of the room, door, window etc.). A positive sign is noted when a swaying, sometimes irregular swaying and even toppling over occurs. The essential feature is that the patient becomes more unsteady with eyes closed. The essential features of the test are as follows:
  1. the subject stands with feet together, eyes open and hands by the sides.
  2. the subject closes the eyes while the examiner observes for a full minute. Romberg's test is positive if the patient falls while the eyes are closed. Swaying is not a positive sign as it shows proprioceptive correction.

CONTACTS AND LOCATIONS:
Overall Officials: Layba Marrium, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shields N. Physiotherapy management of Down syndrome. J Physiother. 2021 Oct;67(4):243-251. doi: 10.1016/j.jphys.2021.08.016. Epub 2021 Sep 10. No abstract available. PMID 34511385